CLINICAL TRIAL: NCT00189345
Title: Randomized, Multicenter, 2-Dose Level. Open-Label, Phase IIa Study With the Intraperitoneally Infused Trifunctional Bispecific Antibody Removab(TM) (Anti-EpCAM x Anti-CD3) to Select the Better Dose Level in Platinum Refractory Epithelial Ovarian Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AGO Study Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGO-OVAR 2.10
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2006-11-08 (Estimated); Status verified 2003-12

CONDITIONS: Ovarian Cancer; Fallopian Tube Neoplasms; Peritoneal Neoplasms
Keywords: Cancer; Cancer alternative therapies; ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms; Neoplasms | interventions — catumaxomab

INTERVENTIONS:
Biological: anti-EpCAM x anti-CD3 (removab)

SUMMARY:
Patients with epithelial ovarian cancer, fallopian tube or peritoneal cancer who receive surgical cytoreduction and platinum/taxane containing chemotherapy have a significant chance of entering complete clinical remission but about 70% will eventually relapse. Many patients respond to additional cytotoxic treatment with partial or complete responses, yet approximately 100% of these patients will ultimately progress. Novel consolidation strategies following treatment for recurrent disease are needed and an immunologic approach is an attractive option.EpCAM is expressed in a large number of epithelial ovarian cancer, fallopian tube or peritoneal cancer tissues. Thus targeting these cancers with an anti-EpCAM antibody is a promising innovative therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

women 18 years and older histologically confirmed epithelial ovarian cancer, cancer of the fallopian tube or peritoneum measurable disease signed and dated informed consent one or two prior chemotherapies, the last platinum containing platinum refractory disease ECOG performance status 0-2

Exclusion Criteria:

acute or chronic infections previous treatment with mouse monoclonal antibodies known or suspected hypersensitivity to removab inadequate renal function inadequate hepatic function ileus cachectic patients

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 44
Dates: Start 2004-05; Study Completion 2005-10

PRIMARY OUTCOMES:
Selection of better dose level based on the confirmed tumor response.

SECONDARY OUTCOMES:
Evaluation of safety and tolerability
Effects of removab(TM)

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Wagner, Prof.Dr., Principal Investigator — AGO Study Group
Locations (1):
- Dept. of Gynecology, University of Marburg, Marburg, Germany

REFERENCES:
- [Derived] Baumann K, Pfisterer J, Wimberger P, Burchardi N, Kurzeder C, du Bois A, Loibl S, Sehouli J, Huober J, Schmalfeldt B, Vergote I, Luck HJ, Wagner U. Intraperitoneal treatment with the trifunctional bispecific antibody Catumaxomab in patients with platinum-resistant epithelial ovarian cancer: a phase IIa study of the AGO Study Group. Gynecol Oncol. 2011 Oct;123(1):27-32. doi: 10.1016/j.ygyno.2011.06.004. Epub 2011 Jul 5. PMID 21733566